CLINICAL TRIAL: NCT06588127
Title: Health Behavior Nudge Strategies for Chronic Disease Patients: the Study of Hypertension and Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lin Han (Other)
Responsible Party: Sponsor-Investigator, Lin Han, prof, LanZhou University
Organization: LanZhou University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 722740872020
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Economics, Behavioral; Hypertension; Type 2 Diabetes Mellitus (T2DM); Self-management Behavior; Health Behavior
MeSH Terms: conditions — Behavior; Hypertension; Diabetes Mellitus, Type 2; Health Behavior

STUDY DESIGN:
Intervention Model Description: Select two communities of comparable size and level, with one community recruiting participants as a control group and the other community recruiting participants as an intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nudge Group (Experimental): The research formed an intervention team comprising 1 project leader, 2 project members, 1 community general practitioner, and 3 community nurses. The project leader oversees the project's progress and quality, while the project members implement specific intervention measures. The community general practitioner addresses the health issues faced by patients in their daily lives, and the nurses communicate with both patients and project team members. The intervention is executed on-site and online, with online efforts primarily utilizing WeChat, a widely used social tool in China. The research will span 6 months, with data collection occurring at baseline, 3, and 6 months.
  Interventions: Behavioral: nudge
- Control Group (No Intervention): According to the Basic Public Health Service Specification of China and the Prevention and Control Management Guidelines for Hypertension and Diabetes in Primary Health care, routine community care for HP and T2DM patients should be conducted, including monitoring blood pressure and blood sugar, follow-up on the health status of patients, and distribution of community health promotion materials.

INTERVENTIONS:
Behavioral: nudge — Nudge interventions are developed based on the scoping review and qualitative research by the research team, which involves commitment (behavioral contracts), norms (case and experience sharing), significance and framing effects (posters, health behavior identification posts), reminders, and incentives (arteriosclerosis detection). The content encompasses diet, physical activity, medication management, self-monitoring, and control of smoking and alcohol. From the viewpoint of bounded rationality in behavioral economics, and drawing on prior research that has pinpointed decision-making biases in patients' self-management behaviors, nudging strategies have been developed to assist individuals in overcoming these biases or to utilize the patterns of these biases to steer them toward making choices that are in line with their health.
  Arms: Nudge Group

SUMMARY:
This study is conducted from the perspective of behavioral economics, where individuals often display bounded rationality in decision-making, opting for habitual choices rather than those most advantageous to themselves. Nudge strategies can utilize individuals' cognitive and motivational shortcomings to influence behavior. Therefore, the study first examines the decision-making biases present in patients with hypertension (HP) and type 2 diabetes mellitus (T2DM) regarding the maintenance of healthy behaviors based on individuals' bounded rationality; subsequently, it develops an intervention program to encourage healthy behaviors in HP and T2DM patients alongside nudge strategies; finally, it assesses the intervention effects of the program on blood pressure, blood glucose, and health behaviors in HP and T2DM patients.

DETAILED DESCRIPTION:
The study was conducted in Lanzhou City, Gansu Province, China. The research selected two communities of similar scale and level, recruiting 133 patients with HP and T2DM. A six-month quasi-experimental study was performed, where the intervention group implemented nudging strategies while the control group received standard community nursing. By measuring the patients' blood pressure and blood glucose levels, and utilizing the Diabetes Self-Care Scale, Hypertension Self-Management Behavior rang Scale，Patient Activation Measure，Short-Form Health Survey, Activity of Daily Living Scale to assess the behavioral changes in both groups, validated the intervention effect of the nudging strategy on the health behaviors of patients with HP and T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Previously diagnosed with hypertension, type 2 diabetes, or hypertension combined with type 2 diabetes
* Able to use mobile phones or other electronic devices
* Informed consent

Exclusion Criteria:

* Patients who are pregnant or breastfeeding;
* Patients with severe diabetes, hypertension complications, or other serious illnesses;
* Patients with hearing or vision impairments;
* Patients with cognitive impairments or mental illnesses;
* Patients with acute complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Self-management behavior | Baseline, 3rd month, 6th month
  The self-management behaviors of T2DM patients were evaluated using the Diabetes Self-Care Scale (DSCS), encompasses six dimensions: dietary control, regular exercise, medication adherence, blood glucose monitoring, foot care, and management of high/low blood sugar, consisting of a total of 26 items rated on a 5-point Likert scale, with higher total scores reflecting greater levels of the behaviors. The self-management behaviors of hypertensive patients were assessed using the Chinese Self-Management Behavior Assessment Scale for Hypertensive Patients, which includes six dimensions and 33 items: exercise management, health monitoring, work and rest management, emotional management, medication management, and dietary management, all rated on a 5-point Likert scale, with a minimum score of 33 and a maximum of 165. The higher scores mean a better outcome. These scales are answered by patients according to their actual situation.

SECONDARY OUTCOMES:
Activity of Daily Living | Baseline, 3rd month, 6th month
  The Barthel Index (BI) is a widely used assessment tool for evaluating Activity of Daily Living (ADL), distinguishing individual self-care abilities based on the score. This score encompasses bowel movements, urination, grooming, eating, toileting, transferring, mobility, dressing, climbing stairs, and bathing, with a maximum score of 100. A score of 100 signifies excellent daily living ability without reliance on others; scores above 60 are classified as good, indicating mild functional impairment but sufficient self-care in daily living; scores between 60 and 41 reflect moderate functional impairment with some assistance required; scores between 40 and 21 denote severe functional impairment with considerable dependence on others; scores below 20 indicate complete disability with total reliance on others for daily living. This measurement is assessed during the interaction between the researcher and the participant.
Life quality | Baseline, 3rd month, 6th month
  The research measured patients quality of life during the study using 12-item short form health survey (SF-12), which is a simplified version of the SF-36, comprising 12 items across 8 domains: Physical Functioning (PF), Role Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). Among these, PF, RP, BP, and GH are classified as physical component summary, while VT, SF, RE, and MH are classified as mental component summary. The standard scoring method was used to calculate the scores of each dimension and the total score was from 0 to 100 points, with a higher score indicating a better quality of life for the individual. The scale is answered by the patient based on their current situation.
Blood pressure(BP) | Baseline, 3rd month, 6th month
  Blood pressure(BP) is recorded in a calm environment by designated community nurses with a standardized electronic blood pressure monitor, precise to 1mmHg.
  Patients are grouped into the community. The measuring instruments must adhere to China metrology certification standards. The measurement methods align with the industry standards of the People's Republic of China - Human Health Monitoring and Human Measurement Methods (WS/T424-2013) requirements.
Blood sugar | Baseline, 3rd month, 6th month
  Blood glucose is a random blood glucose measured by community nurses who gather participants in the community. The instruments must adhere to China metrology certification standards. The measurement methods align with the industry standards of the People's Republic of China - Human Health Monitoring and Human Measurement Methods (WS/T424-2013) requirements.
Body Mass Index(BMI) | Baseline, 3rd month, 6th month
  Patients are grouped in the community and measured by community nurses. The readings for patients' height and weight are documented with height accurate to 0.1cm and weight accurate to 0.1kg. BMI is calculated as weight (kg) / height (m²). The normal value range is 18.5 to 23.9 kg/m², <18.5 kg/m² indicates underweight, BMI ≥ 24 kg/m² indicates overweight, and BMI ≥ 28 kg/m² indicates obesity. All measuring instruments must adhere to China metrology certification standards. The measurement methods align with the industry standards of the People's Republic of China - Human Health Monitoring and Human Measurement Methods (WS/T424-2013) requirements.
Patient Activation Measure | Baseline, 3rd month, 6th month
  The research measured patients enthusiasm for self-management during the study using the Patient Activation Measure (PAM). The scale was developed to assess patients' awareness, knowledge, skills, and confidence in self-managing their diseases. This scale is unidimensional and consists of 13 items, with a Cronbach's α of 0.882. It employs a 5-point Likert scale, where scores range from 0 to 4, representing "not at all suitable for me" to "strongly agree," with higher scores indicating greater positivity. The original total score of the scale ranges from 13 to 52 points. Based on the conversion table provided by the original author, the total score is transformed from 0 to 100 points. A score of ≤47 is classified as low, 47-55.1 as low to moderate, 55.2-67 as moderate, and ≥67.1 as high.The scale is answered by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Fanghong Yan, Principal Investigator
Locations (1):
- School of nursing, Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kullgren JT, Hafez D, Fedewa A, Heisler M. A Scoping Review of Behavioral Economic Interventions for Prevention and Treatment of Type 2 Diabetes Mellitus. Curr Diab Rep. 2017 Sep;17(9):73. doi: 10.1007/s11892-017-0894-z. PMID 28755061
- [Background] Peng G, Yan F, Sun R, Zhang Y, Zhao R, Zhang G, Qiao P, Ma Y, Han L. Self-management behavior strategy based on behavioral economics in patients with hypertension: a scoping review. Transl Behav Med. 2024 Jun 27;14(7):405-416. doi: 10.1093/tbm/ibae018. PMID 38776869
- [Background] Forberger S, Wichmann F, Comito CN. Nudges used to promote physical activity and to reduce sedentary behaviour in the workplace: Results of a scoping review. Prev Med. 2022 Feb;155:106922. doi: 10.1016/j.ypmed.2021.106922. Epub 2021 Dec 18. PMID 34933021
- [Background] Modin D, Johansen ND, Vaduganathan M, Bhatt AS, Lee SG, Claggett BL, Dueger EL, Samson SI, Loiacono MM, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Jean-Marie Martel C, Valentiner-Branth P, Krause TG, Biering-Sorensen T. Effect of Electronic Nudges on Influenza Vaccination Rate in Older Adults With Cardiovascular Disease: Prespecified Analysis of the NUDGE-FLU Trial. Circulation. 2023 May 2;147(18):1345-1354. doi: 10.1161/CIRCULATIONAHA.123.064270. Epub 2023 Mar 5. PMID 36871213
- [Background] Hollands GJ, Shemilt I, Marteau TM, Jebb SA, Kelly MP, Nakamura R, Suhrcke M, Ogilvie D. Altering micro-environments to change population health behaviour: towards an evidence base for choice architecture interventions. BMC Public Health. 2013 Dec 21;13:1218. doi: 10.1186/1471-2458-13-1218. PMID 24359583
- [Background] Shapiro MF, Shu SB, Goldstein NJ, Victor RG, Fox CR, Tseng CH, Vangala S, Mogler BK, Reed SB, Villa E, Escarce JJ. Impact of a Patient-Centered Behavioral Economics Intervention on Hypertension Control in a Highly Disadvantaged Population: a Randomized Trial. J Gen Intern Med. 2020 Jan;35(1):70-78. doi: 10.1007/s11606-019-05269-z. Epub 2019 Sep 12. PMID 31515735
- [Background] Blumenthal-Barby JS, Krieger H. Cognitive biases and heuristics in medical decision making: a critical review using a systematic search strategy. Med Decis Making. 2015 May;35(4):539-57. doi: 10.1177/0272989X14547740. Epub 2014 Aug 21. PMID 25145577